CLINICAL TRIAL: NCT02077595
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Cortical Excitability in the Primary Motor Cortex in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 101-3624B
Record Dates: First submitted 2014-02-11; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Transcutaneous Electrical Nerve Stimulation
Keywords: transcutaneous electrical nerve stimulation; transcranial magnetic stimulation
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 120Hz alternating current stimulation group (Active Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation, TENS
- 5Hz alternating current stimulation group (Active Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation, TENS
- sham alternating current stimulation group (Sham Comparator)
  Interventions: Device: transcutaneous electrical nerve stimulation, TENS

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation, TENS — Then participants will receive stimulation for 20 minutes.

SUMMARY:
Recently, non-invasive brain stimulation has become a powerful tool in both basic research and clinical application. Among several non-invasive brain stimulation techniques, transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS) have received the most attention. About DC stimulation, the change of polarity could modulate the spontaneous neuronal activity and make effect on decision making, language, memory, sensory perception, and pain. In spite of that the concept of transcranial alternating current stimulation (tACS) is not novel, AC is relatively safe compared to DC, and researches have revealed that AC might potentially have the effect on the cortical excitability. However, there are still many areas about AC stimulation which remain unknown, such as mechanism, application, and potential influence on cortical excitability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential | Baseline
  measure of intracortical inhibition on abductor pollicis brevis by single-pulse TMS.
Intracortical inhibition, ICI | Baseline,2 hours, 2.5 hours,and 3 hours
  Measure of changes in intracortical inhibition on abductor pollicis brevis by paired-pulse TMS.
intracortical facilitation, ICF | Baseline,Baseline,2 hours, 2.5 hours,and 3 hours
  Measure of changes in intracortical inhibition on abductor pollicis brevis by paired-pulse TMS.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan